CLINICAL TRIAL: NCT00367614
Title: A Multicenter, Randomized, Open-Label, Single And Multiple Dose Study Of The Pharmacokinetics And Safety of Two Dose Levels of Pantoprazole Sodium Tablets In Adolescents Aged 12 Through 16 Years With A Clinical Daignosis Of GERD.
Brief Title: Study Evaluating Pantoprazole in Adolescents With GERD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3001A3-337
Record Dates: First submitted 2006-08-21; First posted 2006-08-23 (Estimated); Last update posted 2007-12-10 (Estimated); Status verified 2007-12

CONDITIONS: Gastroesophageal Reflux
Keywords: Adolescents; GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Pantoprazole

INTERVENTIONS:
Drug: pantoprazole

SUMMARY:
The purpose of this study is characterize the PK profile of single and multiple doses of pantoprazole in adolescents aged 12 to 16 years with Gastroesophageal Reflux Disease (GERD).

ELIGIBILITY:
Inclusion Criteria:

* 12-16 years old
* clinical diagnosis of GERD
* ability to swallow tablets

Exclusion Criteria:

* GI or malabsorption disorders
* chronic use of warfarin
* positive pregnancy test

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2007-01; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Characterization of the PK profile of single and multiple doses of pantoprazole.

SECONDARY OUTCOMES:
Assess the safety and tolerability of pantoprazole.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer